CLINICAL TRIAL: NCT00818792
Title: A Multicenter, Randomized Trial to Compare Xience and Vision Coronary Stents in the Same Multivessel Patient With Chronic Kidney Disease
Brief Title: Randomized Comparison of xiEnce and visioN Coronary Stents in the sAme muLtivessel Patient With Chronic kiDnEy diSease
Acronym: RENAL-DES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Hospital (Other)
Responsible Party: Principal Investigator, Fabrizio Tomai, MD, FACC, FESC, European Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RENAL-DES
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Kidney Disease; Multivessel Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Drug-eluting stent; Chronic kidney disease; Restenosis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug-eluting stent Xience V (Active Comparator)
  Interventions: Device: Coronary stent
- Bare-metal stent Vision (Active Comparator)
  Interventions: Device: Coronary stent

INTERVENTIONS:
Device: Coronary stent — Comparison of bare-metal stent (Vision) and drug-eluting stent (Xience V)
  Other Names: Bare metal stent Vision; Drug-eluting stent Xience V

SUMMARY:
Percutaneous coronary intervention (PCI) with bare metal stent (BMS) in patients with renal insufficiency has shown unsatisfactory results. Indeed, drug-eluting stents (DES) might reduce the incidence of restenosis and therefore of target lesion revascularization procedures in these patients.

We therefore designed a prospective, randomized, multicenter, not-sponsored study to directly compare the efficacy in the prevention of clinical restenosis of everolimus-eluting stent (Xience V) and bare-metal stent (Vision) (both 2nd-generation DES and BMS, respectively), both implanted in the same patient with multivessel disease and renal insufficiency in order to obviate for the multiple and unpredictable characteristics of this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal insufficiency (creatinine clearance <60 ml/min, in dialysis patients included) with at least two significant (>70%) coronary lesions in two major coronary vessels.

Exclusion Criteria:

* Age >85 years
* left main coronary artery disease
* saphenous vein graft disease
* ST-elevation MI (<3 days)
* coronary vessel diameter <2.5 or > 4 mm
* contraindication to long-term double antiplatelet therapy
* CABG indication by consensus (cardiovascular team)
* severe valvular heart disease
* informed consent not obtained

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Ischemia-driven target vessel revascularization | 9 months

SECONDARY OUTCOMES:
Incidence of death and myocardial infarction | in-hospital, 30 days, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Tomai, MD, Principal Investigator — Department of Cardiovascular Sciences, European Hospital, Rome
Locations (2):
- Italy (2):
  - European Hospital, Rome
  - Azienda Ospedaliera Istituti Ospitalieri di Verona, Verona

REFERENCES:
- [Background] Schiffrin EL, Lipman ML, Mann JF. Chronic kidney disease: effects on the cardiovascular system. Circulation. 2007 Jul 3;116(1):85-97. doi: 10.1161/CIRCULATIONAHA.106.678342. PMID 17606856
- [Background] Tomai F, Reimers B, De Luca L, Galassi AR, Gaspardone A, Ghini AS, Ferrero V, Favero L, Gioffre G, Prati F, Tamburino C, Ribichini F. Head-to-head comparison of sirolimus- and paclitaxel-eluting stent in the same diabetic patient with multiple coronary artery lesions: a prospective, randomized, multicenter study. Diabetes Care. 2008 Jan;31(1):15-9. doi: 10.2337/dc07-1377. Epub 2007 Oct 1. PMID 17909090
- [Derived] Tomai F, Ribichini F, De Luca L, Petrolini A, Ghini AS, Weltert L, Spaccarotella C, Proietti I, Trani C, Nudi F, Pighi M, Vassanelli C. Randomized Comparison of Xience V and Multi-Link Vision Coronary Stents in the Same Multivessel Patient With Chronic Kidney Disease (RENAL-DES) Study. Circulation. 2014 Mar 11;129(10):1104-12. doi: 10.1161/CIRCULATIONAHA.113.005186. Epub 2013 Dec 19. PMID 24357403
- [Derived] Tomai F, Petrolini A, De Luca L, Nudi F, Lanza G, Vassanelli C, Ribichini F. Rationale and design of the Randomized comparison of XiEnce V and Multilink VisioN coronary stents in the sAme muLtivessel patient with chronic kiDnEy disease (RENAL-DES) study. J Cardiovasc Med (Hagerstown). 2010 Apr;11(4):310-7. doi: 10.2459/JCM.0b013e3283347e24. PMID 19924001